CLINICAL TRIAL: NCT05948839
Title: Personalized Brain Functional Sector-guided rTMS Therapy Targeting DMPFC for Treatment-resistant Depression
Brief Title: pBFS Guided rTMS Over DMPFC for Treatment-Resistant Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changping Laboratory (Other)
Collaborators: Hebei Mental Health Center (Unknown); Shandong Daizhuang Hospital (Unknown); West China Hospital (Other); The Second Affiliated Hospital of Xinxiang Medical University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPLMDDDM150
Record Dates: First submitted 2023-06-29; First posted 2023-07-17 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Treatment Resistant Depression; Major Depressive Disorder
Keywords: Treatment Resistant Depression, TRD; Moderate Depression, MDD; personalized neuromodulation; Personalized Brain Functional Sectors
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active rTMS treatment (Experimental): 3 sessions of active rTMS would be delivered to the left DMPFC daily, with a session of 1800 pulse.
  Interventions: Device: active rTMS treatment
- sham control (Sham Comparator): 3 sessions of sham rTMS would be delivered to the left DMPFC daily, with a session of 1800 pulse.
  Interventions: Device: sham rTMS treatment

INTERVENTIONS:
Device: active rTMS treatment — Participants will receive 3 sessions per day of 1800 pulses per session, lasting for 21 days. Individualized targets will be generated using the pBFS method.
  Arms: active rTMS treatment
Device: sham rTMS treatment — The parameters in the sham arms are the same as the active stimulation groups. Stimulation was delivered by the same device as the active group fitted with a sham coil.
  Arms: sham control

SUMMARY:
Investigators aim to evaluate the safety and efficacy of pBFS-guided rTMS therapy targeting DMPFC for patients with treatment-resistant depression

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is an established therapy for treatment-resistant depression. The dorsomedial prefrontal cortex (DMPFC), which serves as a connection intermediary of the aberrant functional network in cognitive control and rumination in depression, has been shown to be highly correlated with disease manifestations and post-treatment improvements through several studies involving neuroimaging and brain injury. Research has shown that the response of DMPFC to rTMS is more subject to improving the dimensions of anxiety and insomnia in depression. Therefore, exploring the novel target DMPFC is also beneficial for distinguishing disease dimensions in the future, thereby enabling personalized treatment and improving clinical treatment efficacy.

After being informed about the study and potential risks. All patients giving written informed consent will undergo a screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requirements will be randomized in a double-blind manner in a 2:1 ratio to the active rTMS group, or sham-control group. Then all participants will undergo a 21-day rTMS modulation and a three- and nine-week follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized/outpatient patients aged 18-65 years (inclusive), male or female.
* Meet the diagnostic criteria of DSM-5(Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) for depression disorder without psychotic symptoms, and currently experiencing a recurrence episode.
* Total HAMD17 score ≥20 and total MADRS score ≥25 before randomization.
* Inadequate response to at least one antidepressant trial of adequate doses and duration.
* A stable antidepressant regimen for at least 4 weeks at a dose not lower than the prescribed range of drug use before randomization.
* Voluntarily participate in the trial and sign informed consent. Able to comply with the planned visit, examination and treatment plan, and other study procedures.

Exclusion Criteria:

* Meet DSM-5 diagnostic criteria for other mental disorders (such as schizophrenia spectrum disorders, bipolar and related disorders, neurodevelopmental disorders, neurocognitive disorders, or depressive disorders due to substances and/or medications, depressive disorders due to other medical problems, etc.);
* Patients with a cardiac pacemaker, cochlear implant, or other metal foreign body and any electronic equipment implanted in the body, patients with claustrophobia and other contraindications to magnetic resonance scanning, and patients with contraindications to rTMS treatment;
* Patients with serious or unstable diseases of the cardiovascular, liver, kidney, blood, endocrine, neurological system, and other systems or organs, especially those with organic brain diseases (such as ischemic stroke, cerebral hemorrhage, brain tumor, etc.) and a history of severe brain trauma as judged by the researcher;
* History of epilepsy (presence of at least 2 uninduced seizures more than 24 hours apart, or diagnosis of the epileptic syndrome, or seizures within the past 12 months); Or currently received medications or other treatments that will lower the seizure threshold;
* History of ECT, rTMS, VNS, DBS, tDCS, light therapy, or other physical therapy related to mental illness within 3 months;
* Currently receiving or planning to start formal cognitive or behavioral therapy, or systemic psychological therapy (interpersonal therapy, dynamic therapy, cognitive behavioral therapy, etc.) during the trial.
* Substance abuse or dependence (including alcohol, drugs, and other psychoactive substances) in the past 1 year;
* Female of childbearing potential who plans to become pregnant during the trial.
* Female that is pregnant or breastfeeding.
* Patients in any clinical trials of other drugs or physical therapy within 1 month before the screening.
* First-degree relatives have bipolar affective disorder.
* There is a significant risk of suicide (MADRS item 10 ≥ 5).
* Difficulty or inability to engage in normal communication, understand or follow instructions, and cooperate with treatment and evaluators.
* Investigators think that was inappropriate to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) scores from baseline to Immediate Post-treatment | Baseline and Day 21(Immediate Post-treatment)]
  The Montgomery-Asberg Depression Rating Scale (MADRS) is a validated instrument stratifying the severity of depressive episodes in adults. The MADRS has an overall score ranging from 0 (no depression) to 60 (worst depression).

SECONDARY OUTCOMES:
Remission and response rates were estimated using Montgomery-Asberg Depression Rating Scale(MADRS) | Baseline, Day 21 (Immediate Post-treatment)
  The response is defined as a symptom improvement of ≥50% and remission is defined as a score ≤10 on MADRS
Remission and response rates were estimated using Hamilton Depression Rating Scale (HAMD-17) | Baseline, Day 21 (Immediate Post-treatment)
  The Hamilton Depression Rating Scale (HAMD) is the most widely used clinician-administered depression assessment scale. The HAMD-17 version consists of 17 items，and has an overall score ranging from 0 (no depression) to 52 (worst depression). Higher scores represent higher depression severity. The response is defined as a symptom improvement of ≥50% and remission is defined as a score ≤7 on HAMD-17
Changes in the MADRS from baseline to each visit | Baseline, Day 21 (Immediate Post-treatment), 3-week Post-treatment, 9-week Post-treatment
  The MADRS has an overall score ranging from 0 (no depression) to 60 (worst depression). Higher scores represent higher depression severity.
Changes in the HAMD-17 from baseline to each visit | Baseline, Day 21 (Immediate Post-treatment), 3-week Post-treatment, 9-week Post-treatment
  The Hamilton Depression Rating Scale (HAMD) is the most widely used clinician-administered depression assessment scale. The HAMD-17 version consists of 17 items，and has an overall score ranging from 0 (no depression) to 52 (worst depression). Higher scores represent higher depression severity.
cognitive changes from baseline to day 21(Immediate Post-treatment) | Baseline, Day 21 (Immediate Post-treatment)
  Cognitive scores are measured using Chinese brief cognitive test (C-BCT), including Digit Symbol Substitution Test (DSST), continuous performance test (CPT), Trail-Making Test (TMT), Digit Span Test (DST)

CONTACTS AND LOCATIONS:
Overall Officials: Hesheng Liu, Ph.D., Study Chair — Changping Laboratory
Locations (3):
- China (3):
  - Hebei Mental Health Center, Baoding, Hebei
  - Shandong Daizhuang Hospital, Jining
  - The Second Affiliated Hospital of Xinxiang Medical University, Xinxiang